CLINICAL TRIAL: NCT01398280
Title: A Single Site Evaluation of the Effect of Topical Application of Aminocaproic Acid (ACA) to Inhibit Kallikrein 5 Serine Protease Activity and Production of LL-37 Cathelicidin Peptide, Biochemical Markers of Rosacea-specific Inflammation.
Brief Title: Effects of Aminocaproic Acid (ACA) on Rosacea-specific Inflammation
Acronym: ACA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tissa Hata, MD, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 100867
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Rosacea
Keywords: Rosacea; Dermatology; UCSD; Skin disease
MeSH Terms: conditions — Rosacea; Skin Diseases | interventions — Aminocaproic Acid; Antibodies, Anticardiolipin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aminocaproic Acid (ACA) (Experimental): Subjects will treat their facial skin twice daily for up to 12 weeks with 5-6 visits and 2 telephone visits. Investigator and subject will be blinded. Tape strip samples will be collected from facial skin at each visit to assess Kallikrein 5 (KLK5) activity.
  Interventions: Drug: Topical aminocaproic acid (ACA) mixed with Vanicream
- Vehicle cream (Placebo Comparator): Subjects will apply vehicle twice daily for up to 12 weeks with 5-6 visits and 2 telephone visits. Investigator and subject will be blinded. Tape strip samples will be collected from facial skin at each visit to assess Kallikrein 5 (KLK5) activity.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: Topical aminocaproic acid (ACA) mixed with Vanicream — 25% Aminocaproic acid cream twice daily for up to 12 weeks.
  Arms: Aminocaproic Acid (ACA)
Drug: Vehicle cream — Vehicle cream moisturizer twice daily for up to 12 weeks
  Arms: Vehicle cream

SUMMARY:
The purpose of this study is to determine the effect of topical aminocaproic acid on the immune system by assessing the levels of antimicrobial peptides in the skin of patients with rosacea. It is hypothesized that aminocaproic acid applied topically will alter the body's immune system in patients with rosacea by inhibiting activation of antimicrobial peptides.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or non-pregnant female, 18 - 70 years of age.
* Subjects willing and able to give informed consent.
* Subjects willing and able to comply with the requirements of the study.
* Subject has the clinical diagnosis of at least mild/moderate papulopustular rosacea (3-20 papulopustules) and at least mild erythema.
* Subject has been on a stable dose for greater than 3 months of medications for treatment of concurrent medical condition (including oral contraceptive pills, vasodilators, adrenergic blocking agents) OR the investigator has determined that the medications are unlikely to affect the patient's rosacea and/or treatment during the study
* Subject is in general good health in the opinion of the investigator.
* Subject has a calculated creatinine clearance 100% of normal range.
* Subject has normal baseline labs or in the opinion of the investigator are values are not clinically significant and would not inhibit the ability to monitor the patient for both safety and efficacy throughout the study.

Exclusion Criteria:

* Subject has a diagnosis of Steroid Rosacea or Pyoderma Faciale (rosacea fulminans)
* Subject has a history of Carcinoid, Pheochromocytoma, Serotonin Syndrome or other systemic flushing causes.
* Subject has used facial topical therapies (OTC drug products or prescription products) for any reason within the prior 28 days
* Subject has used systemic corticosteroid or systemic antibiotics (especially doxycycline, minocycline, tetracycline, metronidazole) within the prior 28 days.
* Subject has had laser or light-based treatment for rosacea within the prior 3 months.
* Subject has had systemic retinoids and retinoid derivatives over the past 6 months
* Subject has an active or recent history of any coagulation (hyper or hypo) disorder, genitourinary bleeding, myopathy, cardiomyopathy, rhabdomyolysis or evidence of clinically significant hepatic disease in the opinion of the investigator,
* Subject is taking any medicines or supplements that interfere with blood clotting such as Coumadin, Plavix, or ASA (>81mg/day).
* Subject has a known hypersensitivity or allergy to aminocaproic acid or components of the vehicle.
* Subject is pregnant or lactating or planning a pregnancy during the duration of the study
* Subject has been treated with another investigational device or drug within 28 days prior to study enrollment or intends to participate in a clinical trial concurrent with this study
* Subject has clinically significant findings, medical history or conditions (other than rosacea), which in the opinion of the Investigator may compromise the study, treatment protocol, or safety of the patient or treatment allocation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tissa Hata, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego Perlman Ambulatory Center, La Jolla, California, United States

REFERENCES:
- [Background] Yamasaki K, Di Nardo A, Bardan A, Murakami M, Ohtake T, Coda A, Dorschner RA, Bonnart C, Descargues P, Hovnanian A, Morhenn VB, Gallo RL. Increased serine protease activity and cathelicidin promotes skin inflammation in rosacea. Nat Med. 2007 Aug;13(8):975-80. doi: 10.1038/nm1616. Epub 2007 Aug 5. PMID 17676051
- [Background] Yamasaki K, Gallo RL. The molecular pathology of rosacea. J Dermatol Sci. 2009 Aug;55(2):77-81. doi: 10.1016/j.jdermsci.2009.04.007. Epub 2009 May 29. PMID 19481425

RESULTS

PARTICIPANT FLOW:
Groups:
- Aminocaproic Acid (ACA): Subjects will treat their facial skin twice daily for up to 12 weeks with 5-6 visits and 2 telephone visits. Investigator and subject will be blinded. Tape strip samples will be collected from facial skin at each visit to assess KLK activity and LL-37 expression.
  Topical aminocaproic acid (ACA) mixed with Vanicream: 25% Aminocaproic acid cream twice daily for up to 12 weeks.
- Vehicle Cream: Subjects will apply vehicle twice daily for up to 12 weeks with 5-6 visits and 2 telephone visits. Investigator and subject will be blinded. Tape strip samples will be collected from facial skin at each visit to assess KLK activity and LL-37 expression.
  Vehicle cream: Vehicle cream moisturizer twice daily for up to 12 weeks
Period: Overall Study
Arm/Group | Aminocaproic Acid (ACA) | Vehicle Cream
Started | 11 | 4
Completed | 7 | 4
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aminocaproic Acid (ACA) | Vehicle Cream | Total
Number analyzed (Participants) | 11 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (18.5) | 63 (5.6) | 55.7 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Kallikrein 5 (KLK5) Protease Activity
Description: Serine protease activity of KLK5 in adult skin from patients with rosacea is measured after treatment with vehicle or aminocaproic acid cream. Protease activity of facial skin surface is monitored using a synthetic fluorogenic trypsin-like proteinase substrate. Protease activity is monitored as an increase of fluorescence (RFU/uL) with SpectraMax GEMINI EM.
Time Frame: Up to 12 weeks
Measure: Mean (Standard Deviation); unit: RFU/uL
Arm/Group | Aminocaproic Acid (ACA) | Vehicle Cream
Number analyzed (Participants) | 7 | 4
RFU/uL | 581.1 (261.0) | 816.5 (422.4)

ADVERSE EVENTS:
Arm/Group | Aminocaproic Acid (ACA) | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/4
Other Adverse Events (participants affected / at risk) | 0/11 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No